CLINICAL TRIAL: NCT00811811
Title: Behavioral Neurocardiac Training With Biofeedback Augments Vagal-Heart Rate Modulation and Baroreflex Sensitivity Among Patients With Hypertension
Brief Title: Behavioral Neurocardiac Training and Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Unilever R&D (Industry)
Responsible Party: Robert P. Nolan/Director Behavioural Cardiology Research Unit, University Health Network
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 04-516-BE
Record Dates: First submitted 2008-12-18; First posted 2008-12-19 (Estimated); Last update posted 2008-12-19 (Estimated); Status verified 2008-12

CONDITIONS: Hypertension
Keywords: Hypertension; Biofeedback; Relaxation training
MeSH Terms: conditions — Hypertension | interventions — Autogenic Training

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Behavioral neurocardiac training
  Interventions: Behavioral: Behavioral neurocardiac training
- 2 (Active Comparator): Autogenic relaxation training
  Interventions: Behavioral: Autogenic relaxation training

INTERVENTIONS:
Behavioral: Behavioral neurocardiac training — 6 training sessions scheduled over 8 weeks
  Arms: 1
Behavioral: Autogenic relaxation training — 6 training sessions scheduled over 8 weeks
  Arms: 2

SUMMARY:
This randomized controlled trial will examine whether behavioral neurocardiac training with heart rate variability biofeedback (BNT) augments reduction in ambulatory daytime and 24-hour SBP, DBP and PP, in comparison to an active control intervention (AC, autogenic relaxation training), among subjects diagnosed with hypertension, and following adjustment for medications. In addition, the independent association between the BNT and AC interventions on vagal-heart rate modulation and baroreflex sensitivity will be evaluated during a standardized assessment protocol of mental stress testing. This study extends a previous trial conducted at the UHN, in which we reported that the biofeedback intervention independently augments vagal-heart rate modulation, while reducing symptoms of stress and depressed mood, among subjects diagnosed with cardiovascular disease. Exploratory features of this trial will examine the association between ambulatory blood pressure, vagal-heart rate modulation, baroreflex sensitivity, and markers of inflammatory activity.

ELIGIBILITY:
Inclusion criteria:

* 35 to 64 years of age
* diagnosis of Grade 1 or 2 hypertension (140-159 mmHg or 160-180 mmHg SBP; or 90-99 or 100-110 mmHg DBP, respectively).
* among subjects not prescribed medication, hypertension confirmed by ambulatory BP monitoring: mean 24-hour SBP > 130 mmHg or DBP > 80 mmHg.
* subjects prescribed antihypertensive pharmacotherapy are required to have a treatment regimen that was unchanged for at least 4 months prior to enrollment.

Exclusion criteria:

* diagnosis of cardiovascular disease, clinically significant arrhythmia, sleep disorder, psychiatric illness (eg. psychosis), alcohol/drug dependence within the previous year, or an inability to comprehend English or French

Ages: 35 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2005-05; Primary Completion 2006-08 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Ambulatory daytime and 24-hour systolic blood pressure, diastolic blood pressure, and pulse pressure. | Baseline and Post-treatment (following 6 treatment sessions scheduled over an 8-week interval)

SECONDARY OUTCOMES:
RR interval, vagal-heart rate modulation (high frequency power in RR interval variability [0.15-0.40 Hz/ms2]) and baroreflex sensitivity | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Robert P Nolan, Ph.D., Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Nolan RP, Floras JS, Harvey PJ, Kamath MV, Picton PE, Chessex C, Hiscock N, Powell J, Catt M, Hendrickx H, Talbot D, Chen MH. Behavioral neurocardiac training in hypertension: a randomized, controlled trial. Hypertension. 2010 Apr;55(4):1033-9. doi: 10.1161/HYPERTENSIONAHA.109.146233. Epub 2010 Mar 1. PMID 20194302